CLINICAL TRIAL: NCT06218537
Title: The Role of oAncreatic Enzyme ReplAcement Therapy (PERT) on Mucosal Visibility Before Upper GI Endoscopy
Acronym: AERATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mihai Ciocirlan, Așsociate Professor of Gastroenterology, Carol Davila University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AERATE
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Upper Gastrointestinal Endoscopy

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated in one of the 2 study groups, using a randomization list.
  The test group - 10 minutes before upper GI endoscopy, patients will drink a solution of 50ml water + 2 capsules of KREON 25000 UI, opened (with minimicrospheres, pellets) + 1.2g sodium bicarbonate, mixed. Adding sodium bicarbonate is necessary to dissolve the minimicrospheres of KREON.
  The control group - 10 minutes before upper GI endoscopy, patients will drink a solution of 50ml water + 1.2g sodium bicarbonate, mixed.
Who Masked: Participant, Investigator
Masking Description: One member of the team will prepare the two solutions, test and control solution, each 50 ml, and will give it to the patient, whithout the patient knowing what solution is. After 10 minutes, the investigator will perform upper GI endoscopy, also without him knowing what solution has been administered to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The test group - 10 minutes before upper GI endoscopy, patients will drink a solution of 50ml water + 2 capsules of KREON 25000 UI, opened (with minimicrospheres, pellets) + 1.2g sodium bicarbonate, mixed. Adding sodium bicarbonate is necessary to dissolve the minimicrospheres of KREON.
  Interventions: Diagnostic Test: Test group
- Control group (Sham Comparator): The control group - 10 minutes before upper GI endoscopy, patients will drink a solution of 50ml water + 1.2g sodium bicarbonate, mixed.
  Interventions: Diagnostic Test: Control group

INTERVENTIONS:
Diagnostic Test: Test group — Contains protease from KREON capsules, activated by adding sodium bicarbonate.
  Arms: Test group
Diagnostic Test: Control group — Contains only sodium bicarbonate.
  Arms: Control group

SUMMARY:
The investigators aim to establish wether the administration of pancreatic enzyme replacement therapy (PERT) improves visibility of the mucosa during upper gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Upper gastrointestinal endoscopy is done "a jeun", without any solid foods at least 8 hours before procedure and no water at least 2 hours before procedure.

Often, the visibility of the mucosa is suboptimal due to presence of saliva which lay on the surface of the gastric mucosa forming small bubbles of foam and also the presence of mucus on the mucosal surface. Current strategies to improve mucosa visibility includes ingestion of simethicone, N-acetyl cysteine (N-ACC) an/or pronase, in different combinations, with 10 to 30 minutes before procedure. There are numerous comparative studies which shows their efficacy [1,2,3,4].

Although the guide of the European Society of Gastrointestinal Endoscopy (ESGE) [5] does not formally recommend these, the United Kingdom and the Australian guidelines do formally recommend them [6].

În România simethicone is available, but not pronase.

Research question of the protocol Does ingestion of a pancreatic protease (KREON 25000 UI) before upper GI endoscopy improves the visibility of the gastric mucosa.

Hypothesis Ingestion of a pancreatic protease (KREON 25000 UI) before upper GI endoscopy improves the visibility score of the gastric mucosa.

ELIGIBILITY:
Inclusion Criteria:

* patient with upper gastrointestinal endoscopy indication, with topical pharyngeal anesthesia
* age above 18 years old
* informed consent

Exclusion Criteria:

* allergy to KREON and/or sodium bicarbonate
* upper gastrointestinal bleeding clinically manifest (hematemesis, melena, hematochesia)
* ingested foreign body
* personal history of esophagectomy, partial or total gastectomy
* absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Crema Stomach Cleaning Score (CSCS) | 2 hours
  The CSCS visibility score [4] will be assessed during upper GI endoscopy. For each of the 3 regions (fornix, gastric body and antrum) the maximum score is 3, so the maximum score is 9. An arbitrary cut-off value of less or equal than 5 for a suboptimal visibility has been chosen and higher than 5 for a satisfactory visibility.

SECONDARY OUTCOMES:
Patient satisfaction score | 2 hours
  Patient satisfaction score assessed by a 10 points (0-10) visual analog scale
Endoscopist satisfaction score | 2 hours
  Endoscopist satisfaction score assessed by a 10 points (0-10) visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- "Agrippa Ionescu" Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuo CH, Sheu BS, Kao AW, Wu CH, Chuang CH. A defoaming agent should be used with pronase premedication to improve visibility in upper gastrointestinal endoscopy. Endoscopy. 2002 Jul;34(7):531-4. doi: 10.1055/s-2002-33220. PMID 12170403
- [Background] Chen HW, Hsu HC, Hsieh TY, Yeh MK, Chang WK. Pre-medication to improve esophagogastroduodenoscopic visibility: a meta-analysis and systemic review. Hepatogastroenterology. 2014 Sep;61(134):1642-8. PMID 25436356
- [Background] Li Y, Du F, Fu D. The effect of using simethicone with or without N-acetylcysteine before gastroscopy: A meta-analysis and systemic review. Saudi J Gastroenterol. 2019 Jul-Aug;25(4):218-228. doi: 10.4103/sjg.SJG_538_18. PMID 31044749
- [Background] Manfredi G, Berte R, Iiritano E, Alicante S, Londoni C, Brambilla G, Romeo S, Menozzi F, Griffanti P, Brandi G, Moreschi O, Pezzilli R, Zullo A, Buscarini E. Premedication with simethicone and N-acetylcysteine for improving mucosal visibility during upper gastrointestinal endoscopy in a Western population. Endosc Int Open. 2021 Feb;9(2):E190-E194. doi: 10.1055/a-1315-0114. Epub 2021 Jan 25. PMID 33532557
- [Background] Bisschops R, Areia M, Coron E, Dobru D, Kaskas B, Kuvaev R, Pech O, Ragunath K, Weusten B, Familiari P, Domagk D, Valori R, Kaminski MF, Spada C, Bretthauer M, Bennett C, Senore C, Dinis-Ribeiro M, Rutter MD. Performance measures for upper gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2016 Sep;48(9):843-64. doi: 10.1055/s-0042-113128. Epub 2016 Aug 22. No abstract available. PMID 27548885
- [Background] Beg S, Ragunath K, Wyman A, Banks M, Trudgill N, Pritchard DM, Riley S, Anderson J, Griffiths H, Bhandari P, Kaye P, Veitch A. Quality standards in upper gastrointestinal endoscopy: a position statement of the British Society of Gastroenterology (BSG) and Association of Upper Gastrointestinal Surgeons of Great Britain and Ireland (AUGIS). Gut. 2017 Nov;66(11):1886-1899. doi: 10.1136/gutjnl-2017-314109. Epub 2017 Aug 18. PMID 28821598